CLINICAL TRIAL: NCT04979182
Title: Somatic and Neurobehavioral Clinical Characterization of Frequent Monogenic Forms of Neurodevelopmental Disorders
Brief Title: Clinical Characterization of Frequent Monogenic Forms of Neurodevelopmental Disorders
Acronym: MONOGENETND
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8209
Record Dates: First submitted 2021-07-16; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-04

CONDITIONS: Neurodevelopmental Disorders
Keywords: Neurodevelopmental disorders; Rare disease; Genetic Diseases; Monogenic syndromes; Intellectual Disability; Autism spectrum disorder; Neurobehavioral Manifestations
MeSH Terms: conditions — Neurodevelopmental Disorders; Rare Diseases; Genetic Diseases, Inborn; Intellectual Disability; Autism Spectrum Disorder; Neurobehavioral Manifestations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective is to constitute a precise and exhaustive collection of clinical data (somatic and neurobehavioral data) of individuals affected by various frequent monogenic forms of neurodevelopmental disorders to better characterize the clinical phenotype of these disorders.

A better knowledge of these manifestations is necessary to improve the management of individuals with these disorders.

The secondary objectives of this research are to inform practitioners, patients and their families about the clinical characteristics of these disorders to better understand their diversity and, finally, to improve their screening and diagnosis. Thus, our study aims at establishing clinical scores, linking genotypes and phenotypes and producing documents for professionals (such as the PNDS (National Diagnostic and Care Protocols))

ELIGIBILITY:
Inclusion criteria:

* Minor patient whose age is ≥ 4 years and ≤18 years
* Major patient with intellectual disability
* Patient treated in a participating center for TND linked to a mutation in one of the genes frequently mutated in this pathology, such as the DYRK1A, KMT2A or other genes;
* Patient having previously been seen in genetic consultation
* Parent (or legal guardian) not having expressed, after information, his opposition to the reuse of his data for the purposes of this research.

Exclusion criteria:

- Parent (or legal guardian) who expressed his opposition to participating in the study.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient treated for TND linked to a mutation in one of the genes frequently mutated in this pathology, such as the DYRK1A, KMT2A or other genes
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Study of clinical profiles associated to different monogenic form of NDD | Files analysed retrospectively from January 01, 2015 to March 31, 2020 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Amélie PITON, MD, Principal Investigator — Service de Génétique Moléculaire Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Génétique Moléculaire Hôpitaux Universitaires de Strasbourg, Strasbourg, France